CLINICAL TRIAL: NCT04372628
Title: Trial of Early Therapies During Non-hospitalized Outpatient Window (TREAT NOW) for COVID-19
Brief Title: Trial of Early Therapies During Non-hospitalized Outpatient Window for COVID-19
Acronym: TREATNOW
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Todd Rice, Associate Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 200827
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Lopinavir; Ritonavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Intervention Model Description: Blinded, multicenter, placebo-controlled randomized clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Lopinavir/Ritonavir tablets or unmatched placebo tablets
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 - Lopinavir/Ritonavir (Active Comparator): Lopinavir/Ritonavir 400 mg/100 mg orally twice daily for twenty-eight doses (Days 1-14)
  Interventions: Drug: Lopinavir/Ritonavir 400 mg/100 mg
- Control Group (Placebo Comparator): Placebo unmatched orally twice daily for 14 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lopinavir/Ritonavir 400 mg/100 mg — Lopinavir/Ritonavir tablets
  Other Names: Kaletra
  Arms: Group 1 - Lopinavir/Ritonavir
Other: Placebo — Unmatched placebo
  Arms: Control Group

SUMMARY:
Blinded, multicenter, placebo-controlled, randomized clinical trial evaluating lopinavir/ritonavir vs placebo in early outpatient treatment of adults with COVID-19

DETAILED DESCRIPTION:
We will conduct an investigator-initiated, multicenter, blinded, placebo-controlled, randomized clinical trial evaluating lopinavir/ritonavir vs placebo for early treatment of adults with COVID-19 in the outpatient setting prior to hospitalization. Patients, treating clinicians, and study personnel will all be blinded to study group assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Laboratory-confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection by reverse transcription polymerase chain reaction (RT-PCR) or other molecular test collected within the past 6 days
3. Current symptoms of acute respiratory infection for ≤6 days, defined as one or more of the following: cough, fever, shortness of breath, chest pain, abdominal pain, nausea/vomiting, diarrhea, body aches, weakness/fatigue.

Exclusion Criteria:

1. Prisoner
2. Pregnancy
3. Breast feeding
4. Two individuals from the same household are not enrolled in the study
5. Unable to randomize within 6 days after onset of acute respiratory infection symptoms
6. Hospitalization within the 6 days prior to randomization
7. Inability to swallow oral medications
8. Refusal or inability to be contacted and participate in daily symptom/safety monitoring in English or Spanish during the two-week follow-up period
9. Previous enrollment in this trial
10. Known severe chronic kidney disease requiring dialysis
11. Known severe liver disease [cirrhosis or >3 times upper limit of normal for aspartate aminotransferase (AST) or alanine aminotransferase (ALT) in medical record if available]
12. Known hepatitis B or hepatitis C infection
13. Known history of jaundice
14. Current heavy alcohol use, defined as 8 drinks or more per week for women or 15 drinks or more per week for men
15. Known seizure disorder
16. Known human immunodeficiency virus (HIV) infection
17. Known history of pancreatitis
18. Known history of prolonged QT interval [Long QT Syndrome, patient report, or corrected QT interval (QTc) >500 milliseconds on most recently available electrocardiogram within the past 2 years]
19. Receipt of >1 dose of lopinavir/ritonavir in the 10 days prior to enrollment
20. Known allergy to lopinavir/ritonavir
21. Currently prescribed (with planned continuation) or planned administration during 14-day study period of medication at high risk for QT prolongation as follows:

    Antiarrhythmics: Amiodarone, disopyramide, dofetilide, dronedarone, flecainide, ibutilide, procainamide, propafenone, quinidine, sotalol Anti-cancer: Arsenic trioxide, oxaliplatin, vandetanib Antidepressants: Amitriptyline, citalopram, escitalopram, imipramine Antimicrobials: azithromycin, ciprofloxacin, clarithromycin, erythromycin, fluconazole, levofloxacin, moxifloxacin, pentamidine, hydroxychloroquine Antipsychotics: haloperidol, chlorpromazine, droperidol, olanzapine, pimozide, quetiapine, thioridazine, risperidone, ziprasidone Others: cilostazol, cimetidine, cisapride, donepezil, methadone, ondansetron, sumatriptan
22. Currently prescribed (with planned continuation) or planned administration during 14-day study period of any of the following medications: alfuzosin, apalutamide, astemizole, ergot-containing medicines (including dihydroergotamine mesylate, ergotamine tartrate, methylergonovine), lomitapide, lovastatin, lurasidone, midazolam, phenobarbital, phenytoin, ranolazine, rifampin, sildenafil, simvastatin, St. John's Wort, terfenadine, triazolam. Patients who are on warfarin or fluticasone will be advised to contact their primary care provider to advise them that they are in the trial and possibly receiving lopinavir/ritonavir which can influence levels of either drug and may require more frequent monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Rice, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (6):
- United States (6):
  - University of Colorado School of Medicine, Aurora, Colorado
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Intermountain, Murray, Utah
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Del Rio C, Malani PN. COVID-19-New Insights on a Rapidly Changing Epidemic. JAMA. 2020 Apr 14;323(14):1339-1340. doi: 10.1001/jama.2020.3072. No abstract available. PMID 32108857
- [Background] Fauci AS, Lane HC, Redfield RR. Covid-19 - Navigating the Uncharted. N Engl J Med. 2020 Mar 26;382(13):1268-1269. doi: 10.1056/NEJMe2002387. Epub 2020 Feb 28. No abstract available. PMID 32109011
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Background] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Background] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Perlman S. Another Decade, Another Coronavirus. N Engl J Med. 2020 Feb 20;382(8):760-762. doi: 10.1056/NEJMe2001126. Epub 2020 Jan 24. No abstract available. PMID 31978944
- [Background] Su S, Wong G, Shi W, Liu J, Lai ACK, Zhou J, Liu W, Bi Y, Gao GF. Epidemiology, Genetic Recombination, and Pathogenesis of Coronaviruses. Trends Microbiol. 2016 Jun;24(6):490-502. doi: 10.1016/j.tim.2016.03.003. Epub 2016 Mar 21. PMID 27012512
- [Background] Cui J, Li F, Shi ZL. Origin and evolution of pathogenic coronaviruses. Nat Rev Microbiol. 2019 Mar;17(3):181-192. doi: 10.1038/s41579-018-0118-9. PMID 30531947
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Background] Cheng PK, Wong DA, Tong LK, Ip SM, Lo AC, Lau CS, Yeung EY, Lim WW. Viral shedding patterns of coronavirus in patients with probable severe acute respiratory syndrome. Lancet. 2004 May 22;363(9422):1699-700. doi: 10.1016/S0140-6736(04)16255-7. PMID 15158632
- [Background] Hui DS, Azhar EI, Kim YJ, Memish ZA, Oh MD, Zumla A. Middle East respiratory syndrome coronavirus: risk factors and determinants of primary, household, and nosocomial transmission. Lancet Infect Dis. 2018 Aug;18(8):e217-e227. doi: 10.1016/S1473-3099(18)30127-0. Epub 2018 Apr 18. PMID 29680581
- [Background] Wang Y, Liu Y, Liu L, Wang X, Luo N, Li L. Clinical Outcomes in 55 Patients With Severe Acute Respiratory Syndrome Coronavirus 2 Who Were Asymptomatic at Hospital Admission in Shenzhen, China. J Infect Dis. 2020 May 11;221(11):1770-1774. doi: 10.1093/infdis/jiaa119. PMID 32179910
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Arentz M, Yim E, Klaff L, Lokhandwala S, Riedo FX, Chong M, Lee M. Characteristics and Outcomes of 21 Critically Ill Patients With COVID-19 in Washington State. JAMA. 2020 Apr 28;323(16):1612-1614. doi: 10.1001/jama.2020.4326. PMID 32191259
- [Background] Wilson N, Kvalsvig A, Barnard LT, Baker MG. Case-Fatality Risk Estimates for COVID-19 Calculated by Using a Lag Time for Fatality. Emerg Infect Dis. 2020 Jun;26(6):1339-1441. doi: 10.3201/eid2606.200320. Epub 2020 Jun 17. PMID 32168463
- [Background] Al-Bari MAA. Targeting endosomal acidification by chloroquine analogs as a promising strategy for the treatment of emerging viral diseases. Pharmacol Res Perspect. 2017 Jan 23;5(1):e00293. doi: 10.1002/prp2.293. eCollection 2017 Feb. PMID 28596841
- [Background] Chu CM, Cheng VC, Hung IF, Wong MM, Chan KH, Chan KS, Kao RY, Poon LL, Wong CL, Guan Y, Peiris JS, Yuen KY; HKU/UCH SARS Study Group. Role of lopinavir/ritonavir in the treatment of SARS: initial virological and clinical findings. Thorax. 2004 Mar;59(3):252-6. doi: 10.1136/thorax.2003.012658. PMID 14985565
- [Background] Chen F, Chan KH, Jiang Y, Kao RY, Lu HT, Fan KW, Cheng VC, Tsui WH, Hung IF, Lee TS, Guan Y, Peiris JS, Yuen KY. In vitro susceptibility of 10 clinical isolates of SARS coronavirus to selected antiviral compounds. J Clin Virol. 2004 Sep;31(1):69-75. doi: 10.1016/j.jcv.2004.03.003. PMID 15288617
- [Background] Wu CY, Jan JT, Ma SH, Kuo CJ, Juan HF, Cheng YS, Hsu HH, Huang HC, Wu D, Brik A, Liang FS, Liu RS, Fang JM, Chen ST, Liang PH, Wong CH. Small molecules targeting severe acute respiratory syndrome human coronavirus. Proc Natl Acad Sci U S A. 2004 Jul 6;101(27):10012-7. doi: 10.1073/pnas.0403596101. Epub 2004 Jun 28. PMID 15226499
- [Background] de Wilde AH, Jochmans D, Posthuma CC, Zevenhoven-Dobbe JC, van Nieuwkoop S, Bestebroer TM, van den Hoogen BG, Neyts J, Snijder EJ. Screening of an FDA-approved compound library identifies four small-molecule inhibitors of Middle East respiratory syndrome coronavirus replication in cell culture. Antimicrob Agents Chemother. 2014 Aug;58(8):4875-84. doi: 10.1128/AAC.03011-14. Epub 2014 May 19. PMID 24841269
- [Background] Chan JF, Yao Y, Yeung ML, Deng W, Bao L, Jia L, Li F, Xiao C, Gao H, Yu P, Cai JP, Chu H, Zhou J, Chen H, Qin C, Yuen KY. Treatment With Lopinavir/Ritonavir or Interferon-beta1b Improves Outcome of MERS-CoV Infection in a Nonhuman Primate Model of Common Marmoset. J Infect Dis. 2015 Dec 15;212(12):1904-13. doi: 10.1093/infdis/jiv392. Epub 2015 Jul 21. PMID 26198719
- [Background] Wang J. Fast Identification of Possible Drug Treatment of Coronavirus Disease-19 (COVID-19) through Computational Drug Repurposing Study. J Chem Inf Model. 2020 Jun 22;60(6):3277-3286. doi: 10.1021/acs.jcim.0c00179. Epub 2020 May 4. PMID 32315171
- [Background] Martinez MA. Compounds with Therapeutic Potential against Novel Respiratory 2019 Coronavirus. Antimicrob Agents Chemother. 2020 Apr 21;64(5):e00399-20. doi: 10.1128/AAC.00399-20. Print 2020 Apr 21. PMID 32152082
- [Background] Kim UJ, Won EJ, Kee SJ, Jung SI, Jang HC. Combination therapy with lopinavir/ritonavir, ribavirin and interferon-alpha for Middle East respiratory syndrome. Antivir Ther. 2016;21(5):455-9. doi: 10.3851/IMP3002. Epub 2015 Oct 22. PMID 26492219
- [Background] Spanakis N, Tsiodras S, Haagmans BL, Raj VS, Pontikis K, Koutsoukou A, Koulouris NG, Osterhaus AD, Koopmans MP, Tsakris A. Virological and serological analysis of a recent Middle East respiratory syndrome coronavirus infection case on a triple combination antiviral regimen. Int J Antimicrob Agents. 2014 Dec;44(6):528-32. doi: 10.1016/j.ijantimicag.2014.07.026. Epub 2014 Sep 18. PMID 25288266
- [Background] Min CK, Cheon S, Ha NY, Sohn KM, Kim Y, Aigerim A, Shin HM, Choi JY, Inn KS, Kim JH, Moon JY, Choi MS, Cho NH, Kim YS. Comparative and kinetic analysis of viral shedding and immunological responses in MERS patients representing a broad spectrum of disease severity. Sci Rep. 2016 May 5;6:25359. doi: 10.1038/srep25359. PMID 27146253
- [Background] Chan JF, Chan KH, Kao RY, To KK, Zheng BJ, Li CP, Li PT, Dai J, Mok FK, Chen H, Hayden FG, Yuen KY. Broad-spectrum antivirals for the emerging Middle East respiratory syndrome coronavirus. J Infect. 2013 Dec;67(6):606-16. doi: 10.1016/j.jinf.2013.09.029. Epub 2013 Oct 3. PMID 24096239
- [Background] Lauer SA, Grantz KH, Bi Q, Jones FK, Zheng Q, Meredith HR, Azman AS, Reich NG, Lessler J. The Incubation Period of Coronavirus Disease 2019 (COVID-19) From Publicly Reported Confirmed Cases: Estimation and Application. Ann Intern Med. 2020 May 5;172(9):577-582. doi: 10.7326/M20-0504. Epub 2020 Mar 10. PMID 32150748
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Gao J, Tian Z, Yang X. Breakthrough: Chloroquine phosphate has shown apparent efficacy in treatment of COVID-19 associated pneumonia in clinical studies. Biosci Trends. 2020 Mar 16;14(1):72-73. doi: 10.5582/bst.2020.01047. Epub 2020 Feb 19. PMID 32074550
- [Background] Sapp JL, Alqarawi W, MacIntyre CJ, Tadros R, Steinberg C, Roberts JD, Laksman Z, Healey JS, Krahn AD. Guidance on Minimizing Risk of Drug-Induced Ventricular Arrhythmia During Treatment of COVID-19: A Statement from the Canadian Heart Rhythm Society. Can J Cardiol. 2020 Jun;36(6):948-951. doi: 10.1016/j.cjca.2020.04.003. Epub 2020 Apr 8. PMID 32299753
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Wang Y, Fan G, Salam A, Horby P, Hayden FG, Chen C, Pan J, Zheng J, Lu B, Guo L, Wang C, Cao B. Comparative Effectiveness of Combined Favipiravir and Oseltamivir Therapy Versus Oseltamivir Monotherapy in Critically Ill Patients With Influenza Virus Infection. J Infect Dis. 2020 Apr 27;221(10):1688-1698. doi: 10.1093/infdis/jiz656. PMID 31822885
- [Derived] Kaizer AM, Shapiro NI, Wild J, Brown SM, Cwik BJ, Hart KW, Jones AE, Pulia MS, Self WH, Smith C, Smith SA, Ng PC, Thompson BT, Rice TW, Lindsell CJ, Ginde AA. Lopinavir/ritonavir for treatment of non-hospitalized patients with COVID-19: a randomized clinical trial. Int J Infect Dis. 2023 Mar;128:223-229. doi: 10.1016/j.ijid.2022.12.028. Epub 2022 Dec 27. PMID 36581186
- [Derived] Kaizer AM, Wild J, Lindsell CJ, Rice TW, Self WH, Brown S, Thompson BT, Hart KW, Smith C, Pulia MS, Shapiro NI, Ginde AA. Trial of Early Antiviral Therapies during Non-hospitalized Outpatient Window (TREAT NOW) for COVID-19: a summary of the protocol and analysis plan for a decentralized randomized controlled trial. Trials. 2022 Apr 8;23(1):273. doi: 10.1186/s13063-022-06213-z. PMID 35395957
- See also: World Health Organization (WHO). WHO R&D Blueprint: informal consultation on prioritization of candidate therapeutic agents for use in novel coronavirus 2019 infection, Geneva, Switzerland, 24 January 2020. [Internet]. [cited 2020 Mar 19] — https://apps.who.int/iris/handle/10665/330680
- See also: Woosley R, Heise C, Gallo T, Tate J, Woosley D, Romero K. www.CredibleMeds.org, QTdrugs ListCredibleMeds [Internet]. [cited 2020 Apr 24] — https://www.crediblemeds.org/
- See also: WHO | Coronavirus disease (COVID-2019) R&D [Internet]. WHO. [cited 2020 Mar 18]; — http://www.who.int/blueprint/priority-diseases/key-action/novel-coronavirus/en/
- See also: Hydroxychloroquine [Internet]. In: LiverTox: Clinical and Research Information on Drug-Induced Liver Injury. Bethesda (MD): National Institute of Diabetes and Digestive and Kidney Diseases; 2012 [cited 2020 Mar 21]. — http://www.ncbi.nlm.nih.gov/books/NBK548738/

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1- Hydroxychloroquine: Hydroxychloroquine 400 mg orally twice daily for two doses (Day 1), then 200 mg twice daily for subsequent eight doses (Day 2-5), then placebo twice daily for subsequent eighteen doses (Day 6-14).
  Arm Terminated 6/22/2020
- Group 2 - Lopinavir/Ritonavir: Lopinavir/Ritonavir 400 mg/100 mg orally twice daily for twenty-eight doses (Days 1-14)
  Lopinavir/Ritonavir 400 mg/100 mg: Lopinavir/Ritonavir tablets
- Placebo Control Group: Placebo Group 1: matched to Hydroxychloroquine orally twice daily for 14 days Placebo Group 2: unmatched orally twice daily for 14 days
Period: Overall Study
Arm/Group | Group 1- Hydroxychloroquine | Group 2 - Lopinavir/Ritonavir | Placebo Control Group
Started | 4 | 221 | 227
Completed | 3 | 216 | 221
Not Completed | 1 | 5 | 6

BASELINE CHARACTERISTICS:
Population: No difference in overall number of baseline participants and those assigned to study arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1- Hydroxychloroquine | Group 2 - Lopinavir/Ritonavir | Placebo Control Group | Total
Number analyzed (Participants) | 4 | 221 | 227 | 452
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 215 | 220 | 439
  >=65 years | 0 | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 129 | 133 | 264
  Male | 2 | 92 | 94 | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 20 | 13 | 34
  Not Hispanic or Latino | 3 | 201 | 213 | 417
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3 | 6
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 0 | 16 | 16 | 32
  White | 3 | 183 | 191 | 377
  More than one race | 0 | 8 | 4 | 12
  Unknown or Not Reported | 1 | 10 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 4 | 221 | 227 | 452

OUTCOME MEASURES:

1. Primary Outcome: Modified COVID Ordinal Outcomes Scale: Study Day 15 (Group 2 and Placebo Control Group)
Description: Improvement of clinical condition of the participant defined by the Modified COVID Ordinal Outcomes Scale (Modified from the COVID-19 WHO ordinal Outcomes score to fit the outpatient setting). This scale reflects a range of participants from dead to not hospitalized and with no limitations to activities of daily living. A score of 1 is "death", 2 is "Hospitalized on mechanical ventilation or extracorporeal membrane oxygenator (ECMO)", 3 is "Hospitalized on supplemental oxygen", 4 is "Hospitalized not on supplemental oxygen", 5 is "Not hospitalized with symptoms and limitation in activity", 6 is "Not hospitalized with symptoms but with no limitation in activity", 7 is "Not hospitalized without symptoms nor limitation in activity". COVID outcomes are more severe at the lower end of the scale and milder at the higher end of the scale for this outpatient trial.
Time Frame: Day 1 to Day 15
Population: Includes all randomized participants, Unknown represents those with no daily surveys submitted over the first 15 study days
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Control Group: Placebo Group 2: unmatched orally twice daily for 14 days
Arm/Group | Group 2 - Lopinavir/Ritonavir | Placebo Control Group
Number analyzed (Participants) | 221 | 227
Participants
  Death | 0 | 0
  Hospitalized on Mechanical Ventilation/ECMO | 1 | 0
  Hospitalized on Supplemental Oxygen | 5 | 4
  Hospitalized, Not on Supplemental Oxygen | 1 | 2
  Not Hospitalized, Symptomatic, Limitations to Daily Activities | 187 | 191
  Not Hospitalized, Symptomatic, No Limitations to Daily Activities | 10 | 14
  Not Hospitalized, No Symptoms, No Limitations to Daily Activities | 12 | 10
  Unknown (no participant response) | 5 | 6

2. Secondary Outcome: Modified COVID Ordinal Outcome Scale: Study Day 8 (Group 2 and Placebo Control Group)
Description: as for outcome 1
Time Frame: on or at Day 8
Population: 41 participants did not complete a survey in Group 2 34 participants did not complete a survey in the Placebo Control Group
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 - Lopinavir/Ritonavir | Placebo Control Group
Number analyzed (Participants) | 221 | 227
Participants
  Death | 0 | 0
  Hospitalized on Mechanical Ventilation/ECMO | 1 | 0
  Hospitalized on Supplemental Oxygen | 2 | 1
  Hospitalized, Not on Supplemental Oxygen | 0 | 0
  Not Hospitalized, Symptomatic, Limitations to Daily Activities | 76 | 61
  Not Hospitalized, Symptomatic, No Limitations to Daily Activities | 28 | 51
  Not Hospitalized, No Symptoms, No Limitations to Daily Activities | 73 | 80
  Unknown (No participant response) | 41 | 34

3. Secondary Outcome: Modified COVID Ordinal Outcome Scale: Study Day 29 (Group 2 and Placebo Control Group)
Description: as for outcome 1
Time Frame: on or at Day 29
Population: 58 participants did not complete a survey in Group 2; 38 participants did not complete a survey in the Placebo Control Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 - Lopinavir/Ritonavir | Placebo Control Group
Number analyzed (Participants) | 221 | 227
Participants
  Death | 1 | 0
  Hospitalized on Supplemental Oxygen | 1 | 0
  Hospitalized, Not on Supplemental Oxygen | 1 | 1
  Not Hospitalized, Symptomatic, Limitations to Daily Activities | 9 | 11
  Not Hospitalized, Symptomatic, No Limitations to Daily Activities | 11 | 16
  Not Hospitalized, No Symptoms, No Limitations to Daily Activities | 140 | 161
  Unknown (no participant response) | 58 | 38

4. Secondary Outcome: Number of Patients Hospitalized: Day 1 to 29 (Group 2 and Placebo Control Group)
Description: Number of patients hospitalized from Day 1 to 29 (Group 2 and Placebo Control Group)
Time Frame: Day 1 to Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 - Lopinavir/Ritonavir | Placebo Control Group
Number analyzed (Participants) | 221 | 227
Participants
  Hospitalized | 7 | 6
  Non-hospitalized | 214 | 221

5. Secondary Outcome: Time to Hospitalization Day 1 to Day 29 (Group 2 and Placebo Control Group)
Description: Number of days from enrollment to hospitalization (Group 2 and Placebo Control Group)
Time Frame: Day 1 to Day 29
Population: Those with a recorded hospitalization
Measure: Median (Full Range); unit: days
Arm/Group | Group 2 - Lopinavir/Ritonavir | Placebo Control Group
Number analyzed (Participants) | 7 | 6
days | 6 [2 to 11] | 7 [3 to 13]

6. Secondary Outcome: Time to Symptom Resolution: Day 1 to Day 29 (Group 2 and Placebo Control Group)
Description: Number of days from enrollment to resolution of COVID-19 symptoms (Group 2 and Placebo Control Group)
Time Frame: Day 1 to Day 29
Population: If a respondent did not report symptoms on any survey (e.g., if they resolved before receiving the medication), they were not included in the time to symptom resolution based on how we worded it in the SAP (i.e., time from medication receipt to resolution)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Group 2 - Lopinavir/Ritonavir | Placebo Control Group
Number analyzed (Participants) | 208 | 221
days | 11 [8 to 29] | 11 [7 to 29]

7. Secondary Outcome: All-cause, All-location Mortality: Day 1 to Day 29 (Group 2 and Placebo Control Group)
Description: Survival status (All-cause, all-location mortality) from Day 1 to Day 29 (Group 2 and Placebo Control Group)
Time Frame: Day 1 to Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 - Lopinavir/Ritonavir | Placebo Control Group
Number analyzed (Participants) | 221 | 227
Participants
  Died | 1 | 0
  Alive | 173 | 195
  Unknown | 47 | 32

8. Secondary Outcome: Oxygen-free Days: Day 1 to Day 29 (Group 2 and Placebo Control Group)
Description: Number of Days without oxygen Day 1 to Day 29 (Group 2 and Placebo Control Group)
Time Frame: Day 1 to Day 29
Population: Participants who never filled out a daily survey were excluded since we could not derive oxygen status. We present the median (IQR), and with almost all participants having no days on supplemental oxygen (or with other outcomes); Median (Q1, Q3) all are 17. 5 participants in Group 2 and 6 participants in the placebo never filled out the daily survey.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Group 2 - Lopinavir/Ritonavir | Placebo Control Group
Number analyzed (Participants) | 221 | 227
days | 17 [17 to 17] | 17 [17 to 17]

9. Secondary Outcome: Fever-free Days: Day 1 to Day 29 (Group 2 and Placebo Control Group)
Description: Number of days without fever from Day 1 to Day 29 (Group 2 and Placebo Control Group)
Time Frame: Day 1 to Day 29
Population: Related to outcome 6, if symptoms resolved before receiving medication they were not included in this outcome. 13 participants in Group 2 and 6 participants in Placebo Control group did not fill out the data relevant to tracking fever-free days.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Group 2 - Lopinavir/Ritonavir | Placebo Control Group
Number analyzed (Participants) | 208 | 221
days | 16 [14 to 17] | 17 [15 to 17]

10. Secondary Outcome: Ventilator-free Days: Day 1 to Day 29 (Group 2 and Placebo Control Group)
Description: Number of days without ventilator use from Day 1 to Day 29 (Group 2 and Placebo Control Group)
Time Frame: Day 1 to Day 29
Population: Related to outcome 8, if no daily surveys were completed, we could not derive ventilation status. We present the median (IQR), and with almost all participants having no days on a ventilator; Median (Q1, Q3) all are 17. There was no data for 5 participants in Group 2 and 6 participants in the Placebo Control Group.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Group 2 - Lopinavir/Ritonavir | Placebo Control Group
Number analyzed (Participants) | 216 | 221
days | 17 [17 to 17] | 17 [17 to 17]

11. Secondary Outcome: ICU-free Days: Day 1 to Day 29 (Group 2 and Placebo Control Group)
Description: Number of days outside the ICU from Day 1 to Day 29 (Group 2 and Placebo Control Group)
Time Frame: Day 1 to Day 29
Population: Related to outcome 8, if no daily surveys were completed, we could not determine ICU-free days. We present the median (IQR), and with almost all participants having no days in the ICU; Median (Q1, Q3) all are 17.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Group 2 - Lopinavir/Ritonavir | Placebo Control Group
Number analyzed (Participants) | 216 | 221
days | 17 [17 to 17] | 17 [17 to 17]

12. Secondary Outcome: Hospital-free Days: Day 1 to Day 29 (Group 2 and Placebo Control Group)
Description: Number of days outside the hospital from Day 1 to Day 29 (Group 2 and Placebo Control Group)
Time Frame: Day 1 to Day 29
Population: Related to outcome 8, if no daily surveys were completed we could not determine ICU-free days. We present the median (IQR), and with almost all participants having no hospitalized days; Median (Q1, Q3) all are 17.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Group 2 - Lopinavir/Ritonavir | Placebo Control Group
Number analyzed (Participants) | 208 | 221
days | 17 [17 to 17] | 17 [17 to 17]

13. Secondary Outcome: Vasopressor-free Days Through Study Day 29 (Group 2 and Placebo Control Group)
Description: Number of vasopressor-free days through Study Day 29 (Group 2 and Placebo Control Group)
Time Frame: Day 1 to Day 29
Population: We present the median (IQR), with almost all participants having vasopressor-free days throughout primary follow-up; Median (Q1, Q3) all are 17.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Group 2 - Lopinavir/Ritonavir | Placebo Control Group
Number analyzed (Participants) | 216 | 221
days | 17 [17 to 17] | 17 [17 to 17]

ADVERSE EVENTS:
Time Frame: Enrollment - Study Day 16 (or 48 hours after completion of the study drug administration) Deaths were observed through day 29 per the secondary outcome Measure 7 specification, but AEs were only collected as AEs through study Day 16.
Description: Adverse Event: Any untoward medical occurrence associated with the use of a drug or a study procedure, whether or not considered drug related. The Investigators determined daily if any adverse events occurred during the period from enrollment through study day 16 (or 48 hours after completion of the study drug administration).
Arm/Group | Group 1- Hydroxychloroquine | Group 2 - Lopinavir/Ritonavir | Placebo Control Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/221 | 0/227
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/221 | 1/227
Other Adverse Events (participants affected / at risk) | 2/4 | 203/221 | 211/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1- Hydroxychloroquine (N=4) | Group 2 - Lopinavir/Ritonavir (N=221) | Placebo Control Group (N=227)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Lung Infection
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Multi-Organ Failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1- Hydroxychloroquine (N=4) | Group 2 - Lopinavir/Ritonavir (N=221) | Placebo Control Group (N=227)
Chest Pain (Cardiac disorders) | 1 (1) | 112 (112) | 119 (119)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 120 (120) | 107 (107)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 160 (160) | 122 (122)
Fever (General disorders) | 1 (1) | 115 (115) | 103 (103)
Nausea (General disorders) | 1 (1) | 141 (141) | 113 (113)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT04372628/Prot_001.pdf
  • Statistical Analysis Plan (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT04372628/SAP_002.pdf
  • Informed Consent Form (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT04372628/ICF_003.pdf